CLINICAL TRIAL: NCT05915377
Title: READI-SET-GO:Researching Efficient Approaches to Delirium Identification-Sustaining Effective Translation to Create Gero Friendly Organizations
Brief Title: Researching Efficient Approaches to Delirium Identification-Sustaining Effective Translation
Acronym: READI-SET-GO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Mount Nittany Medical Center (Unknown); Beth Israel Deaconess Medical Center (Other); Penn State Health Milton S Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Donna Fick, Professor, Penn State University
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 10658578
Record Dates: First submitted 2023-05-11; First posted 2023-06-23 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Delirium; Delirium in Old Age; Delirium With Dementia; Delirium Superimposed on Dementia
Keywords: Delirium; Confusion; Altered Mental Status; Acute Metabolic Encephalopathy; Implementation; Screening; Acute Care; Electronic Health Record
MeSH Terms: conditions — Delirium; Confusion

STUDY DESIGN:
Intervention Model Description: Step Wedge
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Partial masking of outcomes assessors and providers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Readi Set Go Patient Oriented Sample (Experimental): Hospitalized older adults at risk of developing delirium providing informed consent will have the UB-CAM integrated into the electronic health record and RSDA delirium assessments.
  Interventions: Other: READI-SET GO UB-CAM delirium screening into EHR
- Readi Set Go Administrative Sample (Experimental): All patient admitted to the study wards for the duration of the study will have the UB-CAM integrated into the electronic health record
  Interventions: Other: READI-SET GO UB-CAM delirium screening into EHR

INTERVENTIONS:
Other: READI-SET GO UB-CAM delirium screening into EHR — UB-CAM Delirium screening tool integrated into EHR with education on best practices for delirium management

SUMMARY:
The goal of this step-wedge trial is to test the implementation of daily nurse screening for delirium in routine care and its impact on outcomes and complications in hospitalized older adults admitted to 6 general medicine/surgery units at 3 hospitals in Pennsylvania and Massachusetts.

The main question[s] it aims to answer are:

* 1. To test the fidelity, accuracy, and durability of implementing daily nurse screening for delirium using the UB-CAM in routine care.
* 2. To evaluate the impact of UB-CAM delirium screening on patient and care partner centered outcomes assessed at one month follow-up interviews 3. To evaluate the impact of UB-CAM screening on rates of delirium complications (falls, pressure injury, aspiration) and adverse delirium management (psychoactive medication use, restraint use).

Participants (patients) will be assessed for delirium on study days 1, 2 and 3 (or until hospital discharge) and will be asked basic demographics. These patients will be contacted by phone 1 month after enrollment to collect information about inpatient facility use and to administer the Delirium Burden Patient Scale.

Participants (care partners) will be interviewed at the patient's discharge to complete the Alzheimer's Disease-8 scale. These care partners will be contacted by phone 1 month after enrollment to complete the Delirium Burden Caregiver Scale and to complete a Qualitative Interview which includes questions about communication and collaboration.

DETAILED DESCRIPTION:
This study will integrate daily delirium screening using the UB-CAM into routine care for every older adult admitted to 6 acute medical/surgical units at 3 hospitals in 2 states. The investigators will conduct a stepped-wedge implementation design, where UB-CAM screening will be launched at a new unit every 6 months over a 42-month study. The investigators will utilize evidence-based implementation strategies and test fidelity, accuracy, durability, and impact using a combination of: 1) electronically captured outcomes measured in all older patients admitted to the study units (administrative sample), 2) research RSDAs (Investigators will utilize masking by not making these RSDA delirium assessment determinations available to the clinical nurses) coupled with patient and care partner reported outcomes measured in a consented nested sample of older adults on the study units (patient-oriented sample), and 3) qualitative research using focus groups and 1:1 interviews with hospital staff, patients, and family care partners. The investigators propose the following Specific Aims, which will also be assessed in subgroups: older adults with AD/ADRD, those aged 80 and older, and their care partners.

Study Samples and Settings: The study population is hospitalized older adults admitted to 6 general medicine/surgery units at 3 hospitals in Pennsylvania and Massachusetts. There are 2 patient study samples:

Patient-Oriented Sample (N=1050) (Aims 1, 2): A non-randomized sample of patients admitted to the 6 study units will provide informed consent and undergo up to 3 reference standard delirium assessments (RSDAs), which will be used in the Aim 1 accuracy analyses. These patients and their family care partners will also be interviewed by telephone 1 month after hospital discharge to measure outcomes for Aim 2. An average of 1 patient per week per unit will be enrolled, or 25 patients over each 6-month study period. There are 6 units and 7 study periods, yielding a total of 1050 patients. Each patient will contribute at least 1 and up to 3 RSDAs. Based on READI, the investigators anticipate a 25% discharge rate each day, thus day 1 RSDAs will be available on 100% of the sample, day 2 on 75%, and day 3 on 50%, yielding 2362 paired nurse screen-RSDAs for Aim 1. The investigators will take advantage of the large eligible: enroll ratio (at least 10:1) to enrich this population for subgroups of interest. Specifically, The investigators will enroll 300 patients with AD/ADRD, and 250 patients from subgroups, which will enable subset analyses by sex, age 80 and older, and the presence of AD/ADRD. The investigators do this by preferentially approaching persons with AD/ADRD and those 80 and older among our eligible patient list. The MPIs used this strategy in READI, which achieved its targets of 35% AD/ADRD.

Administrative Sample (N=20,000) (Aim 3): This consists of all patients aged 70 and older admitted to the 6 study units throughout the study period. Outcomes for Aim 3 will be obtained from pharmacy data (for antipsychotic use), ICD discharge codes (for aspiration and pressure injury), incident reports (for falls), and hospital orders (for restraint use) via a waiver of informed consent. Based on information provided by our study hospitals (Section 3.3.3), each unit has 25-40 patients (average 30), of which approximately 1/3, or 10, will be aged 70 or older. With average length of stay of 3.5 days, there will be approximately 20 patients aged 70 or older admitted to each study unit each week. This results in 520 patients per unit every 6-month study period, or 21,840 patients over 6 units and 42 months. The investigators conservatively round this number to 20,000 patients. This will provide sufficient sample size to examine rarer outcomes related to both complications and management of delirium. These data will be de-identified and the investigators will not attempt to link it back to the patient-oriented sample.

1. To test the fidelity, accuracy, and durability of implementing daily nurse screening for delirium using the UB-CAM in routine care. Hypothesis: Screening will be performed in over 90% of eligible days after launch and remain over 90% throughout the study period. Accuracy will be improved relative to the pre-screening period. Focus groups with hospital staff will identify impediments and facilitators to inform fidelity, durability, and future implementation efforts. (Patient-oriented Sample, Staff sample)
2. To evaluate the impact of UB-CAM delirium screening on patient and care partner centered outcomes assessed at one month follow-up interviews. Hypothesis: UB-CAM screening will increase Healthy Days at Home (HDAH), decrease delirium-related distress, and improve perceptions of communication and collaboration relative to the pre-screening period. These same trends will be seen in subgroups of persons with AD/ADRD. (Patient-oriented sample).
3. To evaluate the impact of UB-CAM screening on rates of delirium complications (falls, pressure injury, aspiration) and adverse delirium management (psychoactive medication use, restraint use). Hypothesis: UB-CAM screening will reduce delirium-related complications and adverse delirium management, relative to the pre-screening period (Administrative sample).

ELIGIBILITY:
Inclusion Criteria:

* General medicine (hospitalist) service
* Age 70 or older
* Expected hospital length of stay of 3 or more days

Exclusion Criteria:

* Inability to communicate adequately in English
* Admitted for terminal care

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1050 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Aim 1: To Find the Percent Agreement Between the Nurse UB-CAM Screen and the Reference Standard Delirium Assessment (RSDA) | Three consecutive hospital days
  Accuracy is defined as the percent agreement between the nurse UB-CAM screen and the RSDA. While false negatives (low sensitivity) are most concerning since delirium is missed, false positives are problematic as well, as they lead to false labeling and unnecessary workups, which burden both patients and hospital staff. In subset analyses, the investigators will also consider sensitivity (among all RSDA positives) and specificity (among all RSDA negatives). Our sample size of 2360 assessments and target 20% delirium positivity rate (achieved in READI), will allow both analyses of accuracy, and subset analyses of sensitivity and specificity. Since each patient will contribute 1-3 assessments, the investigators will account for clustering in the analysis, as the investigators did in READI.11 Clinician identification of delirium during the "pre" period will be captured by EMR documentation. Absence of such documentation will be considered negative identification.
Aim 2: To Measure Healthy Days at Home (HDAH) as Defined by the Medicare Payment Advisory Commission | One month post-hospital
  Our patient/care partner focus group told us that if hospitalized, their primary goal was to return home as soon as possible, and stay home. Healthy Days at Home (HDAH) is a measure developed in conjunction with the Medicare Payment Advisory Commission and is calculated:
  HDAH = 30 days - (Index hospitalization days + Mortality Days + Skilled Nursing Facility Days + Inpatient Rehabilitation Day + Long Term Hospital Days + Hospital Transfer/Readmission Days + Subsequent Emergency Department Visit Days)
  The investigators will obtain information on hospital length of stay and discharge disposition from the EMR. The investigators will get information on subsequent inpatient facility stays, readmissions, and ED
Aim 3: To Measure Three Complications of Delirium | From hospital admission through discharge, an average of 1 week
  This outcome includes 3 delirium-related adverse events-falls, severe pressure injury, and aspiration pneumonia. Each occurs in 2-4% of all hospital discharges, but much more frequently in patients with delirium (relative risk for falls among delirious patients may be > 20). Each prolongs length of stay, and increases need for post-discharge facility use, patient and care partner distress, and mortality. The investigators will design our UB-CAM app such that positive screens will present management tips that will address preventive strategies to reduce these complications. For instance, if a patient screens positive for delirium, feeding should occur out of bed or with the head of the bed at 90 degrees, reducing risk of aspiration. The investigators will identify these complications using incident reports (falls, pressure injury) and ICD discharge codes for each outcome, plus "not present on admission" to ensure these were not pre-existing conditions.

SECONDARY OUTCOMES:
Aim 1: Fidelity: To Find the Percent of Eligible Days With At Least One Completed Nurse Delirium Screen | From hospital admission through discharge, an average of 1 week
  Intervention fidelity is defined as the percent of eligible days with at least one completed nurse delirium screen. In READI, clinicians completed the UB-CAM screen in 97% of eligible days, but this was not a full-scale implementation. The fidelity outcome will be tracked through our EMR implementation program, which will also generate weekly adherence reports that will be shared with site nurse champions. This outcome will be measured only after implementation of delirium screening. Sustainability will be defined as screening completion rate in the study periods after the initial six-month launch.
Aim 2: Patient/Family Care Partner Distress | One month after hospital discharge
  The investigators will use the recently developed and validated Delirium Burden scales for patients and care partners (DEL-B-P and DEL-B-C), which specifically ask about distressing symptoms and behaviors related to delirium and hospital staff reactions to them. These measures, co-developed by Drs. Marcantonio, Fick and Inouye, were chosen due to their direct relevance to delirium, and the investigators refer to them as distress rather than burden scales based on advice from our focus group. Both the DEL-B-P and DEL-B-C scales consist of 8 items, and can be completed by patients and family care partners in 2-3 minutes.
Aim 3: Rate of Use of Physical Restraints or Use of Antipsychotic Medications | From hospital admission through discharge, an average of 1 week
  This outcome will focus on use of physical restraints, and use of antipsychotic medications for sedation. Physical restraints requiring physician orders occur in approximately 1% of all admissions. Antipsychotic use is more common, with rates of 7% among adults aged 65 and older admitted for non-psychiatric reasons. The investigators will identify use of restraints from physician orders, and new antipsychotic use from electronic medication administration records. This information will be obtained as part of the administrative data from each of the institutions. The investigators will design the UB-CAM app such that positive screens will trigger recommendations against use of restraints and antipsychotics in favor of non-pharmacological behavioral management strategies, and hypothesize that delirium screening will reduce these adverse management strategies.

OTHER OUTCOMES:
Aim 2: Patient/Care Partner Perceptions of Communication, Collaboration (Qualitative) | One month after hospital discharge
  The investigators expect variable degrees of engagement by patients/care partners with our delirium screening program, depending on whether they screen positive for delirium. Therefore, the investigators will first ask whether they were contacted by hospital staff about the results of screening. Based on those responses, the investigators will utilize a semi-structured interview guide to elicit information about the experience including the quality of the communication, and whether this led to distress vs. security. The investigators will also ask care partners whether they were asked to collaborate in the plan of care around delirium. The investigators will analyze these results via qualitative methods

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Fick, PhD, Principal Investigator — Penn State University; Edward R Marcantonio, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Mount Nittany Medical Center, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All data generated in the context of this proposal will be rapidly submitted to appropriate databases for public access as soon as the results are published. The investigators will share a limited data set post grant as appropriate following the NIH recommendations and updated policies. Data sharing will include the use of a data sharing agreement, with de-identification of the data such that no identification of individual persons occurs as per the HIPAA Privacy Rule and all legal and ethical requirements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 1 year of publication of the study results. It will be available indefinitely.
Access Criteria: To be determined at a later date